CLINICAL TRIAL: NCT06797817
Title: Tributyrin Treatment in Mild Alzheimer Disease: Assessment of Butyrate Effects Via the Gut-Brain
Acronym: TRIM-GUT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Pablo Román López, Associate Professor, Dean of the Faculty of Health Sciences, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 066160941-160941-4-824
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease (AD)
Keywords: butyrate; cognitive decline; cytokines; oxidative stress; gut microbiome; tributyrin; alzheimer disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — tributyrin

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial (1:1), parallel, and double-blind will be conducted. This study will adhere to the guidelines outlined by the CONsolidated Standards of Reporting Trials (CONSORT)
Who Masked: Participant, Investigator
Masking Description: The process of random assignment of participants will be carried out using opaque envelopes containing the assignment to the butyrate group (experimental group) and the CG group (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tributyrin (Experimental): Participants will receive 1 capsule per day for 12 weeks. Each capsule contains 450 mg of tributyrins. The capsules will have a gelatin coating. In the market, formulations are available with dosages ranging from 200 to 500 mg.
  Interventions: Dietary Supplement: tributyrin
- Placebo (Placebo Comparator): The placebo will consist of potato starch encapsulated under identical conditions to those used for the tributyrin capsules, ensuring adequate blinding of the study. The administration of the placebo will follow the same protocol as that of the intervention group.

INTERVENTIONS:
Dietary Supplement: tributyrin — Participants will receive 1 capsule per day for 12 weeks. Each capsule contains 450 mg of tributyrins. The capsules will have a gelatin coating. In the market, formulations are available with dosages ranging from 200 to 500 mg.
  Arms: Tributyrin
Other: Placebo — The placebo will consist of potato starch encapsulated under identical conditions to those used for the tributyrin capsules, ensuring adequate blinding of the study.

SUMMARY:
The goal of this clinical trial is to learn if tributyrin can help prevent or mitigate cognitive decline in individuals with mild Alzheimer's disease (AD). The trial will also examine the safety and effects of tributyrin on inflammation and gut microbiota. The main questions it aims to answer are:

Does tributyrin reduce inflammation and neurodegeneration markers? How does tributyrin affect gut microbiota and intestinal permeability? Researchers will compare tributyrin to a placebo (a look-alike substance that contains no active ingredient) to evaluate its effectiveness.

Participants will:

Take tributyrin or a placebo every day for 12 weeks. Undergo assessments of cognitive function, blood markers (such as NfL and pTau217), and gut health.

The findings are expected to provide insight into the potential of tributyrin as a preventive intervention for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with mild AD within the past year (ICD-10: F00.1).
* voluntary consent to participate in the study in accordance with the Declaration of Helsinki.
* not currently enrolled in any other clinical trial that could confound the results.

Exclusion Criteria:

* individuals with other potential causes of dementia, such as a history of severe traumatic brain injury, brain tumours, epilepsy, or central nervous system infections.
* individuals involved in an intervention that interferes with the trial (immunosuppressive drugs, steroids, antibiotics, or received chemotherapy in the month prior to the start of the intervention).
* individuals with gastrointestinal disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Change from Baseline to 12 weeks and 24 weeks
  For cognitive evaluation, the Montreal Cognitive Assessment (MoCA) will be utilized, a widely recognized tool developed to identify mild cognitive impairment. In comparison to the Mini-Mental State Examination (MMSE), MoCA exhibits greater sensitivity, particularly in the early stages of AD, allowing for the detection of deficits in areas such as attention, memory, language, abstraction, and executive functions
  The MoCA is assessed on a scale ranging from 0 to 30, where higher scores reflect superior cognitive performance. A score of 26 or higher is typically regarded as within the normal range, whereas lower scores indicate different levels of cognitive impairment.

SECONDARY OUTCOMES:
Levels of SCFAs (Acetate, Propionate and Butyrate) in faeces | Change from Baseline to 12 weeks and 24 weeks
  To evaluate whether butyrate supplementation promotes increased levels of SCFAs, levels of acetate, propionate and butyrate will be measured. Faecal samples will be collected before, after 12 months, and three months post-intervention. Faecal samples will be collected in a home setting using tubes containing a stabilizing medium. The tubes will be hermetically sealed to minimize the risk of SCFAs volatilization and ensure sample integrity. SCFA levels will be quantified using gas chromatography-mass spectrometry (GC-MS) (Agilent Technologies). The units of measure for SCFAs will be expressed in µmol/g of faeces.
Intestinal permeability | Change from Baseline to 12 weeks and 24 weeks
  Plasma ZO-1, a core tight-junction scaffold protein, will be quantified as its reduction reflects epithelial structural loss; decreased butyrate availability is known to downregulate ZO-1 expression and increase paracellular permeability. To complement this structural indicator, LPS-binding protein (LBP) will be measured as the primary marker of systemic exposure to gut-derived LPS, representing the canonical downstream pathway of barrier dysfunction that activates TLR4-NF-κB signaling implicated in AD-related neuroimmune activation. Intestinal fatty-acid-binding protein 2 (I-FABP2) will also be assessed as a sensitive indicator of enterocyte membrane integrity. Samples will be analyzed by ELISA kits for ZO-1 (Catalog: EEL211), for LBP (Catalog: EH297RB) and for I-FABP2 (Catalog: EHFABP2) from Thermo Fisher (California, USA). The samples will be stored at -80°C until analysis. Protein levels will be measured in pg/mL.
Systemic inflammation | Change from Baseline to 12 weeks and 24 weeks
  Due to butyrate has demonstrated the ability to inhibit pro-inflammatory cytokines while promoting the production of anti-inflammatory cytokines as well as reduce oxidative stress markers. The levels of IL-1β, IL-6 TNF-α, IL-10 cytokines. Blood samples will be collected from participants to assess the mentioned cytokines at baseline, at the end of the 12-week intervention, and three months after its conclusion using ELISA kits following the manufacturer's instructions (Thermo Fisher, California, USA). Blood samples will be collected at three points. After the sample collection, they will be centrifuged at 2000 x g for 15 minutes, the serum will be obtained, and the blood samples will be stored at -80°C for subsequent analysis. Cytokine levels will be quantified in pg/mL.
Serum levels of NfL | Change from baseline to 12 weeks and 24 weeks
  Neurofilament light chain (NfL) will be assessed as a robust indicator of large-caliber axonal injury, commonly elevated in contexts of microglial activation and peripheral inflammatory signaling. Plasma NfL will be quantified using commercial ELISA kits following manufacturer instructions (Catalog. for NfL: BMS2362 from Thermo Fisher. The levels will be quantified in pg/mL.
Serum levels of pTau217 | Change from Baseline to 12 weeks and 24 weeks
  Phosphorylated tau at threonine-217 (pTau217), the most specific peripheral marker of early tauopathy, provides a sensitive molecular readout of abnormal τ-kinase activity, which can be exacerbated by chronic systemic inflammation. pTau217 will be quantified using commercial ELISA kits following manufacturer instructions (Catalog. ab318936 from Abcam, Cambridge, United Kingdom). The levels will be quantified in pg/mL.
Serum levels of Amyloid42/40 ratio | Change from Baseline to 12 weeks and 24 weeks
  The amyloid-β42/amyloid- β40 (Aβ42/40) ratio will be quantified as a proxy of amyloidogenic processing, as peripheral cytokine-driven changes can modulate γ- and β-secretase activity and thereby influence amyloid-β dynamics. Plasma Aβ42/40 ratio will be quantified using commercial ELISA kits following manufacturer instructions (Catalog. for Aβ40: KHB3481 and for Aβ42: KHB3441 from Thermo Fisher, California, USA). The levels will measure in pg/ml.
Composition of Intestinal Microbiota (16S rRNA Gene Sequencing) | Change from Baseline to 12 weeks and 24 weeks
  To explore the influence of tributyrin supplementation on the composition of the intestinal microbiota, 16S rRNA gene sequencing will be performed on fecal samples from participants before, at the end of the supplementation, and three months after its conclusion. Total bacterial DNA from fresh stool samples will be extracted using the Fast DNA Stool Kit (Thermo Fisher Scientific, California, USA). The 16S rRNA gene will be sequenced using universal primers (341F/806R) to target the V3-V4 region, following methods outlined in previous studies. The raw data will be processed with QIIME2 software, and further bioinformatics analysis will be performed using the MicrobiomeAnalyst online platform (https://www.microbiomeanalyst.ca). This will include assessments of alpha and beta diversity, core microbiome analysis, and random forest modeling.
Accuracy in N-back Task (Working Memory) | Change from Baseline to 12 weeks and 24 weeks
  To assess working memory, participants will perform the N-back task (in its 3-4 task versions) using the PEBL (Psychology Experiment Building Language) platform. Performance will be measured by accuracy, calculated as the percentage of correct responses, with higher percentages indicating better working memory performance. Accuracy will be recorded on a scale from 0% to 100%.
Reaction Time in N-back Task (Working Memory) | Change from Baseline to 12 weeks and 24 weeks
  Participants' reaction time during the N-back task will be measured in milliseconds, using the PEBL platform. Shorter reaction times generally indicate more efficient cognitive processing.
Verbal memory by Rey Test | Change from Baseline to 12 weeks and 24 weeks
  A comprehensive assessment of neurocognitive abilities will be conducted using neurocomputational tools through the PEBL (Psychology Experiment Building Language) platform. The Rey Test, administered via PEBL, will be used to evaluate both verbal memory and visual memory, providing an integrated measure of episodic memory. Scores for immediate recall range from 0 to 15, and from 0 to 30 for delayed recall, with higher scores indicating better verbal memory performance.
Visual memory by Rey Test | Change from Baseline to 12 weeks and 24 weeks
  A comprehensive assessment of neurocognitive abilities will be conducted using neurocomputational tools through the PEBL (Psychology Experiment Building Language) platform. The Rey Test, administered via PEBL, will be used to evaluate both verbal memory and visual memory, providing an integrated measure of episodic memory. Visual Memory: The Rey Test, applied through PEBL, will assess immediate recall (scores from 0 to 15) and delayed recall (scores from 0 to 30), with higher scores reflecting better visual memory performance.
Sustained attention by CPT | Change from baseline to 12 weeks and 24 weeks
  The Continuous Performance Test (CPT), administered through the PEBL platform, will be used to assess sustained attention, vigilance, and inhibitory control. Participants must respond to target stimuli while inhibiting responses to non-targets. Performance will be quantified using three indices: (i) reaction time (milliseconds), reflecting processing speed; (ii) omission errors (range 0 to the total number of target trials), indicating failures to detect targets; and (iii) commission errors (range 0 to the total number of non-target trials), reflecting impulsive responses to non-targets. Higher omission and commission scores denote poorer sustained attention and inhibitory control, whereas faster and more stable reaction times reflect better attentional performance.
Reaction time in Stroop Test (Attention) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. The Stroop Test will be applied to examine attention, specifically the ability to inhibit automatic responses and manage attention in the presence of conflicting stimuli. Reaction Time will be measured by reaction time (in milliseconds), with shorter times indicating better cognitive control.
Accuracy in Stroop Test (Attention) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. Accuracy, measured through the Stroop Test will be recorded as the percentage of correct responses, ranging from 0% to 100%, with higher percentages reflecting better performance.
Completion Time in KEFS test (Cognitive flexibility) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. To assess cognitive flexibility, the D-KEFS will be used, measuring the capacity to switch between different strategies and adapt to new demands. Completion Time administered through PEBL will be measured by completion time (in seconds), with shorter times indicating better cognitive flexibility.
Accuracy in KEFS test (Cognitive flexibility) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. To assess cognitive flexibility, the D-KEFS will be used, measuring the capacity to switch between different strategies and adapt to new demands. Accuracy measured through the D-KEFS will be recorded, with higher accuracy reflecting better cognitive flexibility.
Accuracy in Go/No-Go test (Inhibition) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. The Go/No-Go test will evaluate inhibition, measuring the ability to control impulsive responses to certain stimuli. Accuracy will be measured by accuracy (the percentage of correct responses), with scores ranging from 0% to 100%. Higher values indicate better control over inhibition.
Reaction time in Go/No-Go test (Inhibition) | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. The Go/No-Go test will evaluate inhibition, measuring the ability to control impulsive responses to certain stimuli. Reaction time will also be assessed in the Go/No-Go test. Faster responses typically indicate more efficient inhibition of impulses. Reaction time may vary depending on the specific version of the task.
Executive functions and impulsivity | Change from Baseline to 12 weeks and 24 weeks
  To conduct a comprehensive assessment of neurocognitive abilities, neurocomputational tools will be employed through the PEBL (Psychology Experiment Building Language) platform, which offers a variety of tests designed to measure different aspects of cognition. The Cambridge Gambling Test (CGT) will be utilized to assess decision-making and risk-taking behaviours, providing insights into the participants' executive functions and impulsivity. Performance is generally evaluated by accuracy (the percentage of correct choices) and the inclination to take risks, where greater accuracy indicates stronger decision-making skills. Risk-taking behavior is measured by the amount of money wagered, with larger wagers indicating a higher tendency to take risks.
Neuropsychiatric Inventory Questionnaire (NPI-Q) | Change from Baseline to 12 weeks and 24 weeks
  To obtain a comprehensive understanding of the clinical manifestations associated with mild AD, in addition to the neurocognitive tools mentioned, the Neuropsychiatric Inventory Questionnaire (NPI-Q) will be employed. This tool allows for the identification and assessment of the severity of common neuropsychiatric symptoms in this population, such as agitation, depression, anxiety, apathy, and disinhibited behaviors, as well as the level of distress these symptoms cause to caregivers. The severity of each symptom is typically rated on a scale from 0 to 12, with higher scores indicating more severe symptoms. Caregiver distress is measured on a scale from 0 to 5, where higher scores reflect greater distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) due to concerns related to participant privacy, confidentiality, and compliance with applicable data protection regulations. Additionally, the resources required to anonymize and securely distribute the data are not currently available.